CLINICAL TRIAL: NCT04022876
Title: A Phase 1b Study of the Dual MDMX/MDM2 Inhibitor, ALRN-6924, for the Prevention of Chemotherapy-induced Myelosuppression
Brief Title: A Study of ALRN-6924 for the Prevention of Chemotherapy-induced Side Effects (Chemoprotection)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: With a favorable safety profile the difference between treatment groups for the primary composite endpoint was not sufficient to generate statistically significant results with the targeted sample size
Sponsor: Aileron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALRN-6924-1-03
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Non Small Cell Lung Cancer; Small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Carboplatin; Pemetrexed; Topotecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 2 NSCLC: ALRN-6924+Carboplatin+Pemetrexed (Experimental)
  Interventions: Drug: ALRN-6924; Drug: Carboplatin; Drug: Pemetrexed
- Part 2 NSCLC: Placebo+Carboplatin+Pemetrexed (Experimental)
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Placebo
- Part 1 SCLC: ALRN-6924+Topotecan (Experimental)
  Interventions: Drug: ALRN-6924; Drug: Topotecan

INTERVENTIONS:
Drug: ALRN-6924 — ALRN-6924 administered IV on Days 0-2 prior to carboplatin and pemetrexed administered IV on Day 1 of every 21-day cycle.
  Arms: Part 2 NSCLC: ALRN-6924+Carboplatin+Pemetrexed
Drug: Carboplatin — Carboplatin administered IV on Day 1 of every 21-day cycle.
  Arms: Part 2 NSCLC: ALRN-6924+Carboplatin+Pemetrexed; Part 2 NSCLC: Placebo+Carboplatin+Pemetrexed
Drug: Pemetrexed — Pemetrexed administered IV on Day 1 of every 21-day cycle.
  Arms: Part 2 NSCLC: ALRN-6924+Carboplatin+Pemetrexed; Part 2 NSCLC: Placebo+Carboplatin+Pemetrexed
Drug: Placebo — Placebo administered IV on Days 0-2 prior to carboplatin and pemetrexed administered IV on Day 1 of every 21-day cycle.
  Arms: Part 2 NSCLC: Placebo+Carboplatin+Pemetrexed
Drug: ALRN-6924 — ALRN-6924 administered IV on Days 0-4 prior to topotecan administered IV on Days 1-5 of every 21-day cycle.
  Arms: Part 1 SCLC: ALRN-6924+Topotecan
Drug: Topotecan — Topotecan administered IV on Days 1-5 of every 21-day cycle.
  Arms: Part 1 SCLC: ALRN-6924+Topotecan

SUMMARY:
This is a Phase 1b, multicenter, 2-part study of ALRN-6924 for the prevention of chemotherapy-induced side effects.

Part 1 SCLC is an open-label, multicenter study of ALRN-6924 for the prevention of chemotherapy-induced side effects in patients with p53-mutated ED SCLC undergoing 2nd-line treatment with topotecan. (Part 1 has completed enrollment).

Part 2 NSCLC is a randomized, double-blind, placebo-controlled, multicenter study of ALRN-6924 for the prevention of chemotherapy-induced side effects in patients with p53-mutated advanced NSCLC of adenocarcinoma histology receiving 1st-line treatment with carboplatin plus pemetrexed with or without immunotherapy.

DETAILED DESCRIPTION:
During Part 1 SCLC, topotecan will be administered per standard practice on Days 1-5 of 21-day cycles. Patients will be randomized to receive 1 of 2 initial ALRN-6924 dose levels, to be administered prior to each planned topotecan dose. The incidence, severity and duration of hematologic toxicities, including neutropenia, thrombocytopenia, and febrile neutropenia, will be determined. The safety and tolerability of each ALRN-6924 dose level will be assessed during Part 1. ALRN-6924 is given either 24 hr or 6 hr prior to each topotecan administration.

Part 2 NSCLC of the study will be conducted in two stages. In Stage 1, a total of 20 patients will be randomized 1:1 to receive (with or without immunotherapy) either carboplatin plus pemetrexed plus ALRN-6924 or carboplatin plus pemetrexed plus placebo.

During Stage 1 of Part 2 NSCLC, two interim analyses will be conducted after 10 and 20 patients, respectively, have been evaluated. The purpose of the two interim analyses is to confirm safety and exclude futility. In Stage 2 of Part 2 NSCLC, an additional 40 patients will be randomized to treatment as described for Stage 1.

Immunotherapy and/or bevacizumab may be used concurrently with chemotherapy and after completion of 1st-line treatment (i.e., for maintenance purposes) as per local standard of care. Time of administration of immunotherapy and/or bevacizumab relative to chemotherapy will follow local standards of care.

ELIGIBILITY:
Phase 1b, Part 2 NSCLC Inclusion Criteria:

* Histopathological confirmation of Stage IV NSCLC of adenocarcinoma histology. Cytological diagnosis of NSCLC is acceptable if sufficient tumor tissue is available for p53 mutation analysis. FDA approved liquid biopsies are also acceptable.
* Presence of one or more p53 mutations.
* Measurable disease using RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Adequate hematological status.
* Adequate hepatic and renal function.

Phase 1b, Part 2 NSCLC Exclusion Criteria:

* Advanced NSCLC tumors with EGFR mutations or ALK re-arrangement or other actionable genetic aberrations for which an approved targeted treatment is available. Patients who received prior treatment with EGFR or ALK inhibitors or other systemic drugs or immunotherapy for NSCLC are not eligible.
* Patients who are candidates for anti-PD-1 monotherapy in 1st line advanced NSCLC (e.g. tumors with high PD-L1 expression).
* Presence of active central nervous system metastases and/or carcinomatous meningitis.
* Significant weight loss (≥15% body weight) within the 4 weeks prior to enrollment.

Phase 1b, Part 1 SCLC Inclusion Criteria:

* Histopathological confirmation of ED SCLC that has recurred or been refractory to one line of treatment with standard platinum-based chemotherapy or immuno-chemotherapy. Patients who received immunotherapy after platinum-based chemotherapy are eligible.
* Presence of one or more p53 mutations.
* Measurable disease using RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* Adequate hematological status.
* Adequate hepatic and renal function.

Phase 1b, Part 1 SCLC Exclusion Criteria:

* More than one line of prior chemotherapy for ED SCLC (prior immunotherapy is permitted, concurrent with or subsequent to first line chemotherapy).
* Presence of active central nervous system metastases and/or carcinomatous meningitis.
* Significant weight loss (≥15% body weight) within the 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Phase 1b Part 2 NSCLC | Approximately 6 months
  Proportion of completed treatment cycles that are free of Grade ≥ 3 hematological toxicities (including neutropenia, anemia, thrombocytopenia and febrile neutropenia), and free of chemotherapy dose reductions, and free of use of growth factors and transfusions.
Phase 1b Part 1 SCLC | Approximately 19 months
  Proportion of patients with National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3/4 treatment emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (8):
  - Arizona Cancer Center, Kingman, Arizona
  - Mount Sinai Cancer Research Program, Miami, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Regional Medical Oncolgy Center, Wilson, North Carolina
  - Gabrail Cancer Institute, Canton, Ohio
  - OSHU CHO Northwest, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Lung Clinic, Banja Luka
  - Clinical Center University of Sarajevo, Oncology Clinic, Sarajevo
- Germany (4):
  - Charité Comprehensive Cancer Center Benjamin Franklin Hamato, Onkologische, Berlin
  - Universitaetsklinikum Heidelberg Thoraxklinik Heidelberg, Heidelberg
  - LMU Klinikum der Universitaet Muenchen, Respiratory Medicine and Thoracic Oncology, Campus Innenstandt, München
  - München Klinik Neuperlach, Klinik für Hamatologie und Onkologie, Studienburo Neuperlach/Harlaching, München
- Italy (6):
  - Istituto Romagnolo per lo Studio dei Tumori, Dino Amadori, Meldola
  - Azienda Ospedaliero, Universitaria di Modena, Policlinico di Modena, Modena
  - Istituto Nazionale Tumori di Napoli, IRCCS, Fondazione, G. Pascale, Napoli
  - Università degli Studi di Pavia, IRCCS, Fondazione, Policlinico San Matteo, Pavia
  - Azienda Unità Sanitaria Locale della Romagna, Ospedale Santa Maria delle Croci, Ravenna
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Szpital Kliniczny Przemienienia Panskiego, Poznan, Poland
- Serbia (4):
  - CHC Bezanijska Kosa, Belgrade
  - University Clinical Centre of Serbia, Pulmonology Clinic, Belgrade
  - Clinical Centre Nis, Clinic for Pulmonary Diseases, Niš
  - Institute for Pulmonary Diseases of Vojvodina, Novi Sad
- Spain (3):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - MD Anderson Cancer Center, Madrid